CLINICAL TRIAL: NCT04838808
Title: Rivaroxaban in Type 2 Myocardial Infarctions: A Feasibility, Placebo-controlled, Double-blinded, Randomized Controlled Trial
Brief Title: Rivaroxaban in Type 2 Myocardial Infarctions
Acronym: R2MI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00105055
Record Dates: First submitted 2021-03-11; First posted 2021-04-09 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2022-05

CONDITIONS: Type II Myocardial Infarction
Keywords: myocardial injury; Type II myocardial infarction; Anticoagulation
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rivaroxaban (Active Comparator): Rivaroxaban 2.5mg oral twice daily for 90-days
  Interventions: Drug: Rivaroxaban 2.5 MG [Xarelto]
- Placebo (Placebo Comparator): Oral placebo tablet twice daily for 90-days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rivaroxaban 2.5 MG [Xarelto] — Rivaroxaban 2.5mg twice daily for 90-days
  Arms: Rivaroxaban
Drug: Placebo — Placebo tablet twice daily for 90-days
  Arms: Placebo

SUMMARY:
This trial is the pilot phase of a randomized controlled trial to test the feasibility of recruiting patients with a type 2 myocardial infarction and randomizing them to low-dose rivaroxaban to reduce the risk of major cardiovascular events.

DETAILED DESCRIPTION:
This trial is an investigator-initiated prospective, single-center, placebo-controlled, double blinded, pilot randomized controlled trial of low-dose rivaroxaban (2.5mg oral twice daily) for 90-days following a type 2 myocardial infarction. The primary feasibility outcome is time to recruitment of 100 participants, stratified by sex.

ELIGIBILITY:
Inclusion Criteria:

1. Participant age ≥ 65years or >45 years and an additional risk factor (smoking, diabetes mellitus, hypertension, dyslipidemia or known atherosclerotic disease)
2. Rise in troponin level, with one troponin value above the 99th percentile of the upper limit of normal deemed to be due to a type 2 myocardial infarction by the attending team within the past 30 days
3. Alive at the time of hospital discharge

Exclusion Criteria:

1. Current use of anticoagulation
2. Current use of dual antiplatelet therapy
3. Advanced kidney disease (eGFR <15ml/min)
4. Previous hemorrhagic stroke at any time or embolic stroke within the past year
5. Previous life-threatening bleeding event
6. Life expectancy less than one year
7. Anticoagulation recommended conditions - atrial fibrillation, pulmonary embolism, deep vein thrombosis, mechanical heart valves, rheumatic mitral valve disease, left ventricular thrombosis
8. Surgery in the previous 30 days
9. Inability to provide informed consent in English
10. Pregnancy, breastfeeding or child bearing potential

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2023-01-03 (Actual)

PRIMARY OUTCOMES:
Feasibility outcome | Through study completion, estimated at 1-year
  Time to recruitment of 100 participants, stratified by sex.

SECONDARY OUTCOMES:
Number of participants who experience a composite of death, stroke or myocardial infarction | 90-days
  Composite of death, stroke or myocardial infarction
Number of participants who experience major bleeding | 90-days
  Major bleeding as per the International Society on Thrombosis and Haemostasis (ISTH) Fatal bleeding, symptomatic bleeding requiring presentation to an acute care facility or bleeding resulting in transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Graham, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No